CLINICAL TRIAL: NCT06569901
Title: To Strengthen the Patients Hope After Discharge From the Intensive Care Unit - a Stepped Wedge Cluster Randomized Trial
Brief Title: Strengthening Hope After ICU Discharge
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Oslo University Hospital (Other)
Collaborators: Vestre Viken Hospital Trust (Other); Diakonhjemmet Hospital (Other)
Responsible Party: Principal Investigator, Tone Rustøen, Reseacher, Professor, Oslo University Hospital
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: 542348
Record Dates: First submitted 2024-08-15; First posted 2024-08-26 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Critical Care
Keywords: Critical Care; Critical Illness; Critical Care Outcomes; Post-ICU; Hope; Intervention study
MeSH Terms: conditions — Critical Illness

STUDY DESIGN:
Intervention Model Description: After recruitment of 25 participants, they will be randomized into five clusters. One cluster at a time, will cross over to the intervention group. This recruitment period will be repeated three times to include a total of 75 participants. Prior the intervention, participants will receive "care as usual" and serve as controls.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Cluster A (Experimental): Cluster A will participate in the Hope Intervention shortly after randomization. Prior the intervention the participants will serve as controls.
  Interventions: Behavioral: Hope Intervention
- Cluster B (Experimental): Cluster B will participate in the Hope Intervention when Cluster A ends, approximately four weeks after randomization. Prior the intervention the participants will serve as controls.
  Interventions: Behavioral: Hope Intervention
- Cluster C (Experimental): Cluster C will participate in the Hope Intervention when Cluster B ends, approximately eight weeks after randomization. Prior the intervention the participants will serve as controls.
  Interventions: Behavioral: Hope Intervention
- Cluster D (Experimental): Cluster D will participate in the Hope Intervention when Cluster C ends, approximately 12 weeks after randomization. Prior the intervention the participants will serve as controls.
  Interventions: Behavioral: Hope Intervention
- Cluster E (Experimental): Cluster E will participate in the Hope Intervention when Cluster D ends, approximately 16 weeks after randomization. Prior the intervention the participants will serve as controls.
  Interventions: Behavioral: Hope Intervention

INTERVENTIONS:
Behavioral: Hope Intervention — Group meetings after hospital discharge reflecting on themes that may have an impact on hope.
  The Hope Intervention consists of four group meetings and two individual conversations during a four week period.

SUMMARY:
The goal of this clinical trial is to evaluate an interventional program that aims to strengthen hope in intensive care unit (ICU) patients in the rehabilitation phase. The main questions it aims to answer are:

To develop and implement a follow-up service to strengthen hope in ICU patients, and to evaluate the effect on hope in a stepped wedge randomized trial.

To identify possible predictive factors (facilitators and barriers) associated with hope.

Participants will be asked to take part in an ICU follow-up service, a "Hope Intervention" consisting of digital individual- and group conversations. The program will address topics that are important for hope, such as active involvement, social relationships, believes and thoughts of the future.

We will compare the level of hope between participants who have completed the "Hope Intervention" to those that have not yet completed the program.

DETAILED DESCRIPTION:
The ICU patient's situation is challenging as they are acutely ill over a prolonged period of time and receive life sustaining treatment in the ICU.

Having hope and belief in a positive future, even when the prospects of such future are uncertain, may give strength and motivation and possibly improve the outcome in the rehabilitation phase. Hope is scarcely described in ICU patients.

Health care professionals need to learn how to best support ICU patients and promote hope during the rehabilitation period. Therefore, the main aim of the present study is to develop, implement and evaluate a follow up service to former ICU patients to strengthen their hope using a stepped wedge cluster randomized control intervention trial (SW-CRT). The secondary aim is to identify possible predictive factors associated with hope.

The intervention will start after hospital discharge and will be carried out in group sessions.

ELIGIBILITY:
Inclusion Criteria:

* Patients ≥18 years
* ICU patient for > 48 hours
* must be able to communicate verbally just after their ICU stay and be able to handle digital meetings

Exclusion Criteria:

* Patients with severe cognitive impairment
* Do not understand and speak Norwegian
* Patients with major psychiatric challenges, suicidal attempts as a reason for ICU stay
* Age over 85 years.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2024-09-10 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2030-09 (Estimated)

PRIMARY OUTCOMES:
Hope | Baseline and 1,2,3,4 and 5 months after baseline
  Level of hope will be measured by Herth Hope Index (HHI). Baseline is measured after the patient has been discharged from the hospital. The HHI consists of 12 items measuring levels of hope related to cognitive and affective factors. Item scores range from 1 (strongly disagree) to 4 (strongly agree) and the total score ranges from 12 to 48. A high score indicates higher level of hope.

SECONDARY OUTCOMES:
Social Provsion Scale | Baseline and 1,2,3,4 and 5 months after baseline
  Level of social support will be measured by Social Provision Scale (SPS). Baseline is measured after hospital discharge. The SPS consists of 16 assertions about social support that may apply to the individual. Item scores options are; strongly disagree, disagree, agree, and strongly agree.
  The total score ranges from 16-64, and a high score indicates a high level of social support.
Charlson comorbidity Index | Within 2 months after inclucion
  Data on comorbidity will be measured with Charlson comorbidity Index (CCI) , collected from the medical record.
  The CCI categorize the patients' comorbidities and each comorbidity has an associated weight (from 1 to 6). The total scor ranges from 0-37, and the higher the score, the more likely the predicted outcome will result in mortality.
Memorial Symptom Assessment Scale | Baseline and 1,2,3,4 and 5 months after baseline
  Level of symptoms is measured by Memorial Symptom Assessment Scale (MSAS). MSAS consist of 28 predefined symptomes, were 0 indicated not having the symptom and 1 indicates having the symptom. Maximum number of predefined symptoms is 28, and indicates a worse outcome. If the respondent answers "yes" on a symptom, they are asked at what time the symptom occured, and to rate the severity and distress of the symptom using a numeric rating scale from 0 to 10. Zero indicating "not at all" and 10 "very much". A higher score indicates a worse outcome.
  Baseline is measured after hospital discharge.
General Perceived Self-Efficacy Scale | Baseline and 1,2,3,4 and 5 months after baseline
  Level of a general sense of perceived self-efficacy is measured by General Perceived Self-Efficacy Scale (GSE).The short-form scale consists of items, and each item scores on a 4-point scale from 1 (not at all true) to 4 (exactly true). Total score ranges from 5-20, where high scores reflect courage and perseverance and coping both with daily hassles and stressful life events Baseline is measured after hospital discharge.
Cognitive Failure Questionnaire | Baseline and 1,2,3,4 and 5 months after baseline
  Level of cognitive function is measured by the Cognitive Failure Questionnaire (CFQ).
  The questionnaire has five responses from "never" (0) to "very often" (4). A lower score indicates better cognition.
  Baseline is measured after hospital discharge.

CONTACTS AND LOCATIONS:
Overall Officials: Tone Rustøen, PhD, Principal Investigator — Oslo University Hospital
Locations (3):
- Norway (3):
  - Vestre Viken HF, Bærum Hospital, Drammen, Akershus
  - Diakonhjemmet Hospital, Oslo
  - Oslo University Hospital, Oslo

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Herth K. Abbreviated instrument to measure hope: development and psychometric evaluation. J Adv Nurs. 1992 Oct;17(10):1251-9. doi: 10.1111/j.1365-2648.1992.tb01843.x. PMID 1430629
- [Background] Schneeweiss S, Wang PS, Avorn J, Glynn RJ. Improved comorbidity adjustment for predicting mortality in Medicare populations. Health Serv Res. 2003 Aug;38(4):1103-20. doi: 10.1111/1475-6773.00165. PMID 12968819
- [Background] Broadbent DE, Cooper PF, FitzGerald P, Parkes KR. The Cognitive Failures Questionnaire (CFQ) and its correlates. Br J Clin Psychol. 1982 Feb;21(1):1-16. doi: 10.1111/j.2044-8260.1982.tb01421.x. PMID 7126941
- [Background] Russell D, Cutrona CE, Rose J, Yurko K. Social and emotional loneliness: an examination of Weiss's typology of loneliness. J Pers Soc Psychol. 1984 Jun;46(6):1313-21. doi: 10.1037//0022-3514.46.6.1313. PMID 6737214
- [Background] Portenoy RK, Thaler HT, Kornblith AB, Lepore JM, Friedlander-Klar H, Kiyasu E, Sobel K, Coyle N, Kemeny N, Norton L, et al. The Memorial Symptom Assessment Scale: an instrument for the evaluation of symptom prevalence, characteristics and distress. Eur J Cancer. 1994;30A(9):1326-36. doi: 10.1016/0959-8049(94)90182-1. PMID 7999421
- [Background] Dufault K, Martocchio BC. Symposium on compassionate care and the dying experience. Hope: its spheres and dimensions. Nurs Clin North Am. 1985 Jun;20(2):379-91. PMID 3846980